CLINICAL TRIAL: NCT03049371
Title: Thai Red Cross AIDS Research Center
Brief Title: Exploration of the Neo-Vagina Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Thai Red Cross AIDS Research Centre (Other)
Collaborators: amfAR, The Foundation for AIDS Research (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: The EN-V Study
Record Dates: First submitted 2017-01-24; First posted 2017-02-10 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-11

CONDITIONS: HIV Infections; Transgender Women
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- sample size 100 (Other): 24 post-op and 100 pre- non- and post-op TGW Study participants need to be of Thai nationality, at least 18 years old, male at birth and self-identify as post-op TGW for participation in study. Signed informed consent is required for study participation
  Interventions: Other: No Intervention for both groups

INTERVENTIONS:
Other: No Intervention for both groups — No Intervention for both groups However, computer-administered questionnaire will collect quantitative demographic information and details about surgical history, neovaginal health, neovaginal practices, and sexual behavior including neovaginal intercourse and drug use history from each participant

SUMMARY:
The current study will explore behavioral, surgical and biological neovaginal and rectal HIV transmission risks and feasibility of collection of blood and ano-genital samples (rectal, genital and neo-vaginal, including urine) for microbiological, immunological and cytological characterization in the context of antiretroviral chemoprophylaxis for the prevention of HIV infection in TGW. This includes the feasibility of home self-collection of ano-genital samples prior to habitual cleansing of the anatomical collection site.

DETAILED DESCRIPTION:
A computer-administered questionnaire will collect quantitative demographic information and details about surgical history, neovaginal health, neovaginal practices, and sexual behavior including neovaginal intercourse and drug use history from each participant. The questionnaire can be completed online from any location or at the study clinic and will take about 15-20 minutes.

ELIGIBILITY:
Inclusion Criteria:

Participants will be recruited through existing social networks among TGW and from the Thai Red Cross Anonymous and Tangerine Clinics providing HIV testing, care and treatment services. TGW attending clinic services will be offered enrollment in the study. Particular attention will be paid to offering enrollment to those attending HIV treatment and care services. The current study offers medical evaluation and a range of laboratory testing specific to the health of TGW, which may be of interest and beneficial to them. At the same time, the study may benefit from their participation.

Exclusion Criteria:

not TGW

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2013-01 (Actual); Primary Completion 2019-05 (Actual); Study Completion 2022-11 (Actual)

PRIMARY OUTCOMES:
important information regarding the willingness and obstacles for TGW to come forward for neo-vaginal and rectal HIV and STI evaluation, a computer-administered questionnaire. | 5 years
  A computer-administered questionnaire will collect quantitative demographic information and details about surgical history, neo-vaginal health, neo vaginal practices, and sexual behavior including neo-vaginal intercourse and drug use history from each participant. The questionnaire can be completed online from any location or at the study clinic and will take 15-20 minutes.

CONTACTS AND LOCATIONS:
Overall Officials: Frits van Griensven, PhD, MPH, Principal Investigator — The Thai Red Cross AIDS Research Centre
Locations (1):
- The Thai Red Cross AIDS Research Centre, Pathum Wan, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No